CLINICAL TRIAL: NCT01666444
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Study of VTX-2337 in Combination With Pegylated Liposomal Doxorubicin (PLD) in Patients With Recurrent or Persistent Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: VTX-2337 and Pegylated Liposomal Doxorubicin (PLD) in Patients With Recurrent or Persistent Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GOG-3003
Record Dates: First submitted 2012-08-10; First posted 2012-08-16 (Estimated); Results first posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: recurrent epithelial ovarian cancer; recurrent fallopian tube cancer; recurrent primary peritoneal cavity cancer; ovarian serous cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian mucinous cystadenocarcinoma; ovarian undifferentiated adenocarcinoma; ovarian clear cell cystadenocarcinoma; ovarian mixed epithelial carcinoma; Brenner tumor
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Brenner Tumor | interventions — liposomal doxorubicin; VTX-2337

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PLD 40 mg/m2 plus VTX-2337 (Experimental): The dosing schedule will be be based on a 28-day cycle. The starting dose schedule is PLD on Day 1 plus VTX-2337 on Day 3, Day 10, and Day 17 for the first 4 cycles. Starting with cycle 5, the dose regimen will be PLD on Day 1 plus VTX-2337 on Day 3 only, without additional doses of VTX-2337 on Days 10 and Day 17.
  Interventions: Drug: pegylated liposomal doxorubicin (PLD); Drug: VTX-2337
- PLD 40 mg/m2 plus placebo (Active Comparator): The dosing schedule will be based on a 28-day cycle. The starting dose schedule is PLD on Day 1 plus placebo on Day 3, Day 10, and Day 17 for the first 4 cycles. Starting with cycle 5, the dose regimen will be PLD on Day 1 plus placebo on Day 3 only.
  Interventions: Drug: pegylated liposomal doxorubicin (PLD); Drug: Placebo

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin (PLD)
  Other Names: Doxil; Lipodox
Drug: VTX-2337 — TLR8 Agonist
  Arms: PLD 40 mg/m2 plus VTX-2337
Drug: Placebo
  Arms: PLD 40 mg/m2 plus placebo

SUMMARY:
The purpose of this study is to compare the overall survival of patients treated with VTX-2337 + pegylated liposomal doxorubicin (PLD) versus those treated with PLD alone in women with recurrent or persistent, epithelial ovarian, fallopian tube or primary peritoneal cancer.

VTX-2337, a small molecule agonist of Toll-like Receptor 8 (TLR8), activates multiple components of the innate immune system and is being developed as a novel therapeutic agent for use in oncology. Experimental data obtained in an animal model of ovarian cancer supports the combination of VTX-2337 with PLD. In this model, the combination of VTX-2337 and PLD resulted in a significant reduction in tumor growth compared to either agent alone and an increase in the number of T lymphocytes infiltrating the tumor. The combination of PLD and VTX-2337 has been tested in a small number of women with ovarian cancer in a Phase 1b study and appears to be generally well-tolerated.

DETAILED DESCRIPTION:
OBJECTIVES

Primary Objectives:

* To compare the overall survival (OS) of patients treated with VTX-2337 + PLD versus those treated with PLD alone in women with recurrent or persistent, epithelial ovarian, fallopian tube or primary peritoneal cancer.
* To compare the progression-free survival (PFS) between the two treatment groups using Immune-Related Response Evaluation Criteria in Solid Tumors (irRECIST).

Secondary Objectives:

* To compare the progression-free survival (PFS) between the two treatment groups using Response Evaluation Criteria In Solid Tumors (RECIST 1.1).
* To compare the nature, frequency and severity of drug-related adverse events (AEs) between the two treatment groups.

Exploratory Objectives:

* To compare the best overall response rate (ORR) and duration of response (based on the probability of being in response function [PBRF]) between the two treatment groups using irRECIST and RECIST 1.1.
* To compare the disease control rate (DCR) between the two treatment groups using irRECIST and RECIST 1.1.
* To assess the impact of immune status and response on the clinical effects (OS, PFS, DCR, ORR, PBRF, AEs) of study treatment.
* To assess the effect of TLR8 polymorphisms and BRCA1/BRCA2 mutations on the clinical effects (OS, PFS, DCR, ORR, PBRF, AEs) of study treatment.
* To assess the effect of immune cell subsets, as measured by immunohistochemistry and micro RNA in primary tumor tissue (e.g. immune score), on the clinical effects (OS, PFS, DCR, ORR, PBRF, AEs) of study treatment.
* To assess whether the presence of autoantibodies to tumor-derived proteins are predictive of the clinical effects (OS, PFS, DCR, ORR, PBRF, AEs) of study treatment.

OUTLINE:

This is Phase 2 multicenter clinical study to evaluate the efficacy and safety of the combination of VTX-2337 + PLD compared to PLD + Placebo.

The dosing schedule will be the same for both treatment arms, and will be based on a 28-day cycle. The starting dose schedule is PLD on Day 1 plus VTX-2337 or placebo on Day 3, Day 10, and Day 17 for the first 4 cycles. Starting with cycle 5, the dose regimen will be PLD on Day 1 plus VTX-2337 or placebo on Day 3.

Blood samples are collected periodically during cycle 1 for pharmacodynamics, pharmacogenomics, and other research studies.

Patients will receive therapy until disease progression based on Immune-Related RECIST or until adverse effects prohibit further therapy. Following treatment completion, all patients will be followed with physical exams and histories every three months for the first two years, and then every six months for the next three years, and then

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have recurrent or persistent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma.
2. Patients with the following histologic cell types are eligible: serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial adenocarcinoma, transitional cell carcinoma, malignant Brenner's tumor or adenocarcinoma not otherwise specified.
3. Patient must have measurable disease as defined by RECIST 1.1.
4. Patients must have received treatment with a platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin or another organoplatinum compound. This initial treatment may have included intraperitoneal therapy, consolidation, non-cytotoxic agents or extended therapy administered after surgical or non-surgical assessment.

   Patients are allowed to receive, but are not required to receive, one additional cytotoxic regimen for management of recurrent or persistent disease.

   Patients are allowed to have received, but are not required to have received, biologic/targeted therapy (e.g., bevacizumab and/or PARP inhibitor) as part of their primary treatment regimen or for management of recurrent or persistent disease.
5. Patients must have platinum-resistant disease, defined as having a platinum-free interval (PFI) of < 12 months after first- or second-line platinum-based chemotherapy, or having disease progression while receiving second-line platinum-based chemotherapy.
6. Patients must have adequate bone marrow, renal, hepatic, and neurologic functions as defined by the following:

   * Bone marrow function: absolute neutrophil count (ANC) ≥ 1,500/mm3. This ANC cannot have been induced or supported by granulocyte colony stimulating factors. Platelets ≥ 100,000/mm3. Hemoglobin ≥ 9 g/dL.
   * Renal function: creatinine ≤ 1.5 x institutional upper limit normal (ULN).
   * Hepatic function: bilirubin < 1.2 mg/dL, SGOT (AST) and SGPT (ALT) ≤ 3.0 x ULN and alkaline phosphatase ≤ 2.5 x ULN.
7. Patients must have recovered from effects of recent surgery, radiotherapy or chemotherapy:

   * Patients should be free of active infection requiring parenteral antibiotics.
   * Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration. Continuation of hormone replacement therapy is permitted.
   * Any other prior therapy directed at the malignant tumor, including chemotherapy, biologic/targeted agents and immunologic agents, must be discontinued at least three weeks prior to registration.
   * Any prior radiation therapy must be completed at least four weeks prior to registration.
8. Patients must have a GOG performance status of 0 or 1.
9. Patients of childbearing potential must have a negative pregnancy test prior to the study entry and be practicing an effective form of contraception. If applicable, patients must discontinue breastfeeding prior to study entry.
10. Patients must meet the entry requirements and undergo the baseline procedures.
11. Patients must have signed an IRB-approved informed consent form and authorization permitting release of personal health information.

Exclusion Criteria:

1. Patients who have had treatment with VTX-2337, doxorubicin, PLD, or any other anthracycline.
2. Patients who have received an investigational agent < 30 days prior to registration.
3. Patients who have received oral or parenteral corticosteroids < 2 weeks prior to registration or who require ongoing systemic immunosuppressive therapy for any reason.
4. Patients with active autoimmune disease. "Active" refers to any condition currently requiring therapy. Examples of autoimmune disease include systemic lupus erythematosus, multiple sclerosis, inflammatory bowel disease and rheumatoid arthritis.
5. Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of the other malignancy being present within the last three years.
6. Patients who have received prior radiotherapy OTHER THAN for the treatment of ovarian, fallopian tube or primary peritoneal cancer within the last three years are excluded.
7. Patients who have received prior chemotherapy OTHER THAN for the treatment of ovarian, fallopian tube or primary peritoneal cancer within the last three years are excluded.
8. Patients with history or evidence upon physical examination of CNS disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of treatment on this study.
9. Patients with clinically significant cardiovascular disease.
10. Patients who are pregnant or nursing.
11. Patients under the age of 18.
12. Patients with clinical symptoms or signs of gastrointestinal obstruction and/or who require parenteral hydration or nutrition.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2012-10-31 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley J. Monk, MD, Study Chair — St. Joseph's Hospital and Medical Center, Phoenix AZ; Amar Patel, MD, Study Director — Celgene
Locations (136):
- United States (136):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Winthrop P. Rockefeller Cancer Institute - University of Arkansas, Little Rock, Arkansas
  - Providence Saint Joseph Medical Center, Burbank, California
  - Kaiser Permanente Medical Center, Hayward, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Kaiser Permanente Medical Center, Oakland, California
  - Kaiser Permanente Medical Center, Roseville, California
  - Sutter Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center, San Francisco, California
  - Kaiser Permanente Medical Center, San Jose, California
  - Kaiser Permanente Medical Center, Santa Clara, California
  - Kaiser Permanente Medical Center, South San Francisco, California
  - Stanford University School of Medicine, Stanford, California
  - Kaiser Permanente Medical Center, Vallejo, California
  - Kaiser Permanente Medical Center, Walnut Creek, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - St. Francis Hospital and Medical Center, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale - New Haven Hospital, New Haven, Connecticut
  - MD Anderson Cancer Center - Orlando, Orlando, Florida
  - Women's Cancer Associates, St. Petersburg, Florida
  - Northside Hospital, Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Central Georgia Gynecologic Oncology, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - St. Joseph's - Candler Gynecologic Oncology, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Northwestern University - Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Sudarshan K. Sharma, MD, LTD, Hinsdale, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - St. Vincent Gynecologic Oncology, Indianapolis, Indiana
  - McFarland Clinic, Ames, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Westwood, Kansas
  - Maine Medical Partners Women's Health, Scarborough, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins Medical Institution, Baltimore, Maryland
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - University of Massachusetts Memorial Healthcare, Worcester, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Karmanos Cancer Institute - Wayne State University, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Grand Rapids Clinical Oncology, Grand Rapids, Michigan
  - Saint Mary's Health Care, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Gynecologic Oncology of West Michigan, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Mercy Health Partners - Mercy Campus, Muskegon, Michigan
  - Reed City Hospital - Spectrum Health, Reed City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Minnesota Oncology Coon Rapids Clinic, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Metro Minnesota Clinical Oncology Program, Saint Louis Park, Minnesota
  - Park Nicollet Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - Minnesota Oncology Hematology - St. Paul Cancer Center, Saint Paul, Minnesota
  - Woodbury Clinic - CornerStone Medical Specialty Centre, Woodbury, Minnesota
  - St. Dominic-Jackson Memorial Hospital, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center - University of Missouri, Columbia, Missouri
  - Women's Cancer Care Center of Nevada, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Southwest Gynecologic Oncology Associates, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center, Las Cruces, New Mexico
  - Women's Cancer Care Associates, Albany, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Monter Cancer Center, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - NYU Langone Medical Center - Cancer Institute, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Gynecologic Oncology of Central New York - SUNY Upstate, Syracuse, New York
  - Hope Women's Cancer Center, Asheville, North Carolina
  - Alamance Regional Cancer Center, Burlington, North Carolina
  - Carolinas Medical Center / Levine Cancer Institute, Charlotte, North Carolina
  - Carolinas Medical Center - Northeast, Concord, North Carolina
  - Wake Forest University Health Science, Winston-Salem, North Carolina
  - Summa Health System, Akron, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Fairview Hospital Moll Pavilion Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Women's Cancer Center at Kettering Medical Center, Kettering, Ohio
  - Hillcrest Hospital - Cleveland Clinic, Mayfield Heights, Ohio
  - Lake University Seidman Cancer Center, Mentor, Ohio
  - Peggy and Charles Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Abington Memorial Hospital; Hanjani Institute for Gynecologic Oncology, Abington, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Hillman Cancer Center - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital (McGlinn Family Regional Cancer Center), West Reading, Pennsylvania
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Bon Secours St. Francis Hospital, Greenville, South Carolina
  - Gibbs Cancer Center, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - Mid Atlantic Pelvic Surgery Associates, Annandale, Virginia
  - Virginia Gynecology Oncology, Richmond, Virginia
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - Pacific Gynecology Specialists, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Northwest Hospital - UW Medicine, Seattle, Washington
  - Women's Cancer Care of Seattle, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Green Bay Oncology at St. Vincent's Hospital, Green Bay, Wisconsin
  - St Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology at St. Mary's Hospital, Green Bay, Wisconsin
  - University of Wisconsin-Madison, Madison, Wisconsin
  - Holy Family Memorial Medical Center, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Aurora St. Luke's Medical Center Gynecologic Oncology, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin

REFERENCES:
- [Derived] Newhouse R, Nelissen E, El-Shakankery KH, Rogozinska E, Bain E, Veiga S, Morrison J. Pegylated liposomal doxorubicin for relapsed epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Jul 5;7(7):CD006910. doi: 10.1002/14651858.CD006910.pub3. PMID 37407274
- [Derived] Monk BJ, Brady MF, Aghajanian C, Lankes HA, Rizack T, Leach J, Fowler JM, Higgins R, Hanjani P, Morgan M, Edwards R, Bradley W, Kolevska T, Foukas P, Swisher EM, Anderson KS, Gottardo R, Bryan JK, Newkirk M, Manjarrez KL, Mannel RS, Hershberg RM, Coukos G. A phase 2, randomized, double-blind, placebo- controlled study of chemo-immunotherapy combination using motolimod with pegylated liposomal doxorubicin in recurrent or persistent ovarian cancer: a Gynecologic Oncology Group partners study. Ann Oncol. 2017 May 1;28(5):996-1004. doi: 10.1093/annonc/mdx049. PMID 28453702

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was initiated on 2012-Aug-13 and terminated on 2014-Apr-11. During this time, 297 patients were enrolled.
Pre-assignment Details: Prior to enrollment and treatment assignment, a completed eligibility checklist was electronically checked for completeness and compliance with eligibility criteria. Prior to treatment assignment, patients were stratified by prior platinum free interval (<6 months or >6-12 months) and performance status (0 or 1). Treatments were double-blinded.
Groups:
- Pegylated Liposomal Doxorubicin (PLD) + Placebo: Pegylated Liposomal Doxorubicin (PLD) 40 mg/m2 plus placebo
- Pegylated Liposomal Doxorubicin (PLD)+VTX-2337 (VTX): Pegylated Liposomal Doxorubicin (PLD) 40 mg/m2 plus VTX-2337 3.0 mg/m2
Period: Overall Study
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) + Placebo | Pegylated Liposomal Doxorubicin (PLD)+VTX-2337 (VTX)
Started | 149 | 148
Completed | 147 | 147
Not Completed | 2 | 1
Not completed — Did not initiate treatment | 2 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) + Placebo | Pegylated Liposomal Doxorubicin (PLD)+VTX-2337 (VTX) | Total
Number analyzed (Participants) | 149 | 148 | 297
Age, Continuous [Median (Full Range); unit: years] | 61.6 [29.7 to 91.1] | 63.5 [39.6 to 84.8] | 62.7 [29.7 to 91.1]
Age, Customized [Count of Participants; unit: Participants]
  <40 years | 4 | 1 | 5
  40-49 years | 22 | 11 | 33
  50-59 years | 39 | 42 | 81
  60-69 years | 50 | 51 | 101
  70-79 years | 31 | 38 | 69
  > 79 years | 3 | 5 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 148 | 297
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 143 | 145 | 288
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 141 | 137 | 278
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status is used to describe a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.).
  The scale ranges from 0 to 5:
  0 = Fully active, no restrictions;
  1. = Restricted activity but ambulatory, able to carry out work of a light nature;
  2. = Ambulatory and capable of all self-care but unable to carry out work activities;
  3. = Limited self-care, confined to bed or chair more than 50% of waking hours;
  4. = Completely disabled, no self-care, confined to bed or chair;
  5. = Dead
  Participants
    0 = Fully active, no restrictions | 104 | 105 | 209
    1=Restricted activity;ambulatory;can do light work | 45 | 43 | 88
Prior Platinum-Free Interval as per Case Report Forms [Count of Participants; unit: Participants]
  <= 6 months | 79 | 72 | 151
  > 6 months | 70 | 76 | 146
Prior Chemotherapy Regimens [Count of Participants; unit: Participants]
  1 | 81 | 69 | 150
  2 | 64 | 74 | 138
  3 | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Comparison of duration of survival between the 2 treatment groups
Time Frame: Survival is measured from date of enrollment and randomization on the study until death from any cause, or if alive at last contact, date of last contact.
Population: All enrolled patients
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) + Placebo | Pegylated Liposomal Doxorubicin (PLD)+VTX-2337 (VTX)
Number analyzed (Participants) | 149 | 148
days | 574 [242 to 1141] | 552 [240 to 869]
Statistical Analysis 1: Comparison: Pegylated Liposomal Doxorubicin (PLD) + Placebo vs Pegylated Liposomal Doxorubicin (PLD)+VTX-2337 (VTX); The null hypothesis is that the hazards of death are equal for both treatment groups. The primary assessment of this hypothesis was done with a stratified logrank test and the study was to be considered sufficiently mature to assess this hypothesis when at least 211 deaths had occurred among all individuals enrolled. Type I error was to be set to 0.08 for a one-sided test and the power for detecting a 30% reduction in the hazard (hazard ratio=0.70) due to VTX-2337 was 88.2%; Test type: Superiority or Other; p = 0.923, Log Rank — P-value is for a one-sided hypothesis test; The logrank test is stratified for platinum-free interval (<= 6 months vs > 6 months), and performance status (0 vs 1); Hazard Ratio (HR) = 1.22, 92% CI 1-sided [upper limit 1.48] — Treatment Hazard ratio for overall survival (PLD+VTX relative to PLD+placebo). Survival is measured from date of enrollment and randomization on the study until death from any cause, or date of last contact

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Comparison of PFS between the 2 treatment groups
Time Frame: Progression-free survival is measured from enrollment and randomization on the study until first indication of progression based on irRECIST criteria or death from any cause, or if progression-free at last contact, the date of last disease assessment.
Population: All enrolled patients.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) + Placebo | Pegylated Liposomal Doxorubicin (PLD)+VTX-2337 (VTX)
Number analyzed (Participants) | 149 | 148
days | 159 [87 to 351] | 147 [85 to 267]
Statistical Analysis 1: Comparison: Pegylated Liposomal Doxorubicin (PLD) + Placebo vs Pegylated Liposomal Doxorubicin (PLD)+VTX-2337 (VTX); The null hypothesis is that the hazards of first progression or death are equal for both treatment groups. The primary assessment was to use a stratified logrank test and the study was to be considered sufficiently mature when survival is mature for analysis. Type I error was to be set to 0.02 for a one-sided test and the power for detecting a 31% reduction in the hazard (hazard ratio=0.69) due to VTX-2337 was expected to be approximately 83%; Test type: Superiority or Other; p = 0.943, Log Rank — P-value is for a one-sided hypothesis test; The logrank test is stratified for platinum-free interval (<= 6 months vs > 6 months), and performance status (0 vs 1); Hazard Ratio (HR) = 1.21, 98% CI 1-sided [upper limit 1.56]

3. Secondary Outcome: Frequency and Severity of Adverse Events (AEs)
Description: An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. An AE can be unfavorable and unintended sign, symptom, or disease which is temporally associated with the use of investigational product (IP), whether or not considered related to the IP. A serious AE = an AE occurring at any dose that: • Results in death • Is life- threatening • Requires or prolongs existing inpatient hospitalization • Results in persistent or significant disability/incapacity • Is a congenital anomaly/birth defect; • Constitutes an important medical event. The Investigator assessed the relationship of each AE to IP and graded the severity according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0: Grade (GR) 1 = Mild; asymptomatic or mild symptoms; GR 2 = Moderate (minimal, local or noninvasive intervention indicated); GR 3 = Severe or medically significant; GR 4 = Life-threatening; GR 5 = Death
Time Frame: Assessed during each cycle of therapy and within 30 days after the last cycle of therapy
Population: All patients who initiated study treatment. There were 147 patients who initiated treatment on each arm.
Measure: Number; unit: participants
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) + Placebo | Pegylated Liposomal Doxorubicin (PLD)+VTX-2337 (VTX)
Number analyzed (Participants) | 147 | 147
participants
  Grade 1 | 8 | 3
  Grade 2 | 40 | 44
  Grade 3 | 83 | 90
  Grade 4 | 10 | 3
  Grade 5 | 6 | 7

ADVERSE EVENTS:
Time Frame: Adverse Event assessments began with initiation of any study treatment up until 30 days following the last cycle of treatment.
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) + Placebo | Pegylated Liposomal Doxorubicin (PLD)+VTX-2337 (VTX)
Serious Adverse Events (participants affected / at risk) | 30/147 | 36/147
Other Adverse Events (participants affected / at risk) | 147/147 | 147/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegylated Liposomal Doxorubicin (PLD) + Placebo (N=147) | Pegylated Liposomal Doxorubicin (PLD)+VTX-2337 (VTX) (N=147)
Anemia (Blood and lymphatic system disorders) | 3 | 2
Atrial Fibrillation (Cardiac disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 4
Vomiting (Gastrointestinal disorders) | 5 | 7
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Bloating (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 3 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 6
Mucositis Oral (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 8 | 9
Esophageal Ulcer (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 1
Pain (General disorders) | 0 | 2
Malaise (General disorders) | 1 | 1
Injection Site Reaction (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Edema Limbs (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 4
Death Nos (General disorders) | 0 | 1
Fever (General disorders) | 1 | 3
Chills (General disorders) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 5 | 1
Lung Infection (Infections and infestations) | 0 | 1
Cecal Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 2
Enterocolitis Infectious (Infections and infestations) | 1 | 0
Biliary Tract Infection (Infections and infestations) | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0
Lymphocyte Count Decreased (Investigations) | 1 | 0
Inr Increased (Investigations) | 0 | 1
Creatinine Increased (Investigations) | 4 | 0
Neutrophil Count Decreased (Investigations) | 1 | 2
Blood Bilirubin Increased (Investigations) | 0 | 1
White Blood Cell Decreased (Investigations) | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 1
Alkaline Phosphatase Increased (Investigations) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 3
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Stroke (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Cognitive Disturbance (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 2
Respiratory, Thoracic And Mediastinal Disorders - (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thromboembolic Event (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegylated Liposomal Doxorubicin (PLD) + Placebo (N=147) | Pegylated Liposomal Doxorubicin (PLD)+VTX-2337 (VTX) (N=147)
Anemia (Blood and lymphatic system disorders) | 103 | 105
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 2
Ventricular Tachycardia (Cardiac disorders) | 1 | 0
Sinus Bradycardia (Cardiac disorders) | 1 | 2
Palpitations (Cardiac disorders) | 8 | 6
Heart Failure (Cardiac disorders) | 0 | 1
Atrial Flutter (Cardiac disorders) | 0 | 1
Cardiac Disorders - Other (Cardiac disorders) | 1 | 1
Pericardial Effusion (Cardiac disorders) | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 11 | 6
Chest Pain - Cardiac (Cardiac disorders) | 1 | 1
Middle Ear Inflammation (Ear and labyrinth disorders) | 1 | 0
Ear And Labyrinth Disorders - Other (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 4 | 5
Hearing Impaired (Ear and labyrinth disorders) | 0 | 4
Ear Pain (Ear and labyrinth disorders) | 3 | 1
External Ear Inflammation (Ear and labyrinth disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Eye Disorders - Other (Eye disorders) | 3 | 1
Watering Eyes (Eye disorders) | 2 | 2
Flashing Lights (Eye disorders) | 1 | 2
Eye Pain (Eye disorders) | 0 | 3
Cataract (Eye disorders) | 4 | 0
Conjunctivitis (Eye disorders) | 2 | 1
Blurred Vision (Eye disorders) | 6 | 5
Dry Eye (Eye disorders) | 3 | 2
Floaters (Eye disorders) | 1 | 2
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 17 | 12
Dyspepsia (Gastrointestinal disorders) | 13 | 22
Duodenal Obstruction (Gastrointestinal disorders) | 2 | 0
Dry Mouth (Gastrointestinal disorders) | 10 | 7
Colonic Obstruction (Gastrointestinal disorders) | 4 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 75 | 79
Diarrhea (Gastrointestinal disorders) | 52 | 45
Cheilitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 48 | 70
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Bloating (Gastrointestinal disorders) | 26 | 24
Small Intestinal Perforation (Gastrointestinal disorders) | 1 | 0
Stomach Pain (Gastrointestinal disorders) | 7 | 2
Small Intestinal Obstruction (Gastrointestinal disorders) | 13 | 12
Anal Hemorrhage (Gastrointestinal disorders) | 1 | 1
Anal Mucositis (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 54 | 61
Periodontal Disease (Gastrointestinal disorders) | 1 | 0
Rectal Hemorrhage (Gastrointestinal disorders) | 1 | 3
Obstruction Gastric (Gastrointestinal disorders) | 1 | 0
Small Intestinal Mucositis (Gastrointestinal disorders) | 0 | 2
Mucositis Oral (Gastrointestinal disorders) | 57 | 56
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 3 | 5
Anal Pain (Gastrointestinal disorders) | 0 | 1
Oral Hemorrhage (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 3 | 5
Ileal Obstruction (Gastrointestinal disorders) | 1 | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 2 | 1
Gastric Hemorrhage (Gastrointestinal disorders) | 1 | 0
Oral Pain (Gastrointestinal disorders) | 10 | 10
Abdominal Distension (Gastrointestinal disorders) | 15 | 15
Nausea (Gastrointestinal disorders) | 93 | 97
Gastroparesis (Gastrointestinal disorders) | 2 | 1
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 12 | 15
Rectal Pain (Gastrointestinal disorders) | 1 | 1
Lip Pain (Gastrointestinal disorders) | 0 | 1
Esophageal Ulcer (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 7 | 2
Fecal Incontinence (Gastrointestinal disorders) | 0 | 1
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 3
Ascites (Gastrointestinal disorders) | 15 | 8
Toothache (Gastrointestinal disorders) | 3 | 3
Esophageal Pain (Gastrointestinal disorders) | 1 | 5
Dental Caries (Gastrointestinal disorders) | 3 | 0
Flatulence (Gastrointestinal disorders) | 6 | 6
Gastritis (Gastrointestinal disorders) | 2 | 2
General Disorders And Administration Site Conditio (General disorders) | 3 | 7
Pain (General disorders) | 23 | 26
Malaise (General disorders) | 7 | 6
Localized Edema (General disorders) | 2 | 1
Irritability (General disorders) | 0 | 1
Injection Site Reaction (General disorders) | 13 | 107
Infusion Site Extravasation (General disorders) | 2 | 0
Flu Like Symptoms (General disorders) | 8 | 45
Edema Trunk (General disorders) | 2 | 1
Non-Cardiac Chest Pain (General disorders) | 6 | 3
Edema Limbs (General disorders) | 19 | 37
Facial Pain (General disorders) | 2 | 1
Edema Face (General disorders) | 0 | 1
Fatigue (General disorders) | 109 | 127
Fever (General disorders) | 19 | 70
Gait Disturbance (General disorders) | 2 | 2
Chills (General disorders) | 25 | 92
Infusion Related Reaction (General disorders) | 1 | 5
Hepatobiliary Disorders - Other (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Anaphylaxis (Immune system disorders) | 1 | 0
Allergic Reaction (Immune system disorders) | 4 | 4
Cytokine Release Syndrome (Immune system disorders) | 2 | 24
Immune System Disorders - Other (Immune system disorders) | 1 | 1
Infections And Infestations - Other (Infections and infestations) | 4 | 2
Wound Infection (Infections and infestations) | 1 | 0
Upper Respiratory Infection (Infections and infestations) | 3 | 4
Tooth Infection (Infections and infestations) | 1 | 1
Stoma Site Infection (Infections and infestations) | 1 | 0
Vulval Infection (Infections and infestations) | 2 | 0
Soft Tissue Infection (Infections and infestations) | 1 | 1
Skin Infection (Infections and infestations) | 6 | 16
Sinusitis (Infections and infestations) | 6 | 4
Sepsis (Infections and infestations) | 1 | 0
Salivary Gland Infection (Infections and infestations) | 0 | 1
Rash Pustular (Infections and infestations) | 1 | 1
Peripheral Nerve Infection (Infections and infestations) | 1 | 0
Papulopustular Rash (Infections and infestations) | 3 | 2
Nail Infection (Infections and infestations) | 1 | 2
Mucosal Infection (Infections and infestations) | 3 | 2
Lymph Gland Infection (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 2 | 3
Eye Infection (Infections and infestations) | 1 | 0
Device Related Infection (Infections and infestations) | 1 | 1
Gum Infection (Infections and infestations) | 0 | 2
Vaginal Infection (Infections and infestations) | 4 | 2
Urinary Tract Infection (Infections and infestations) | 12 | 12
Catheter Related Infection (Infections and infestations) | 1 | 0
Joint Infection (Infections and infestations) | 1 | 0
Bronchial Infection (Infections and infestations) | 3 | 0
Bone Infection (Infections and infestations) | 1 | 0
Bladder Infection (Infections and infestations) | 3 | 1
Lip Infection (Infections and infestations) | 0 | 3
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Vascular Access Complication (Injury, poisoning and procedural complications) | 2 | 0
Vaginal Anastomotic Leak (Injury, poisoning and procedural complications) | 0 | 1
Urostomy Obstruction (Injury, poisoning and procedural complications) | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 2 | 0
Radiation Recall Reaction (Dermatologic) (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 3 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 7
Wound Complication (Injury, poisoning and procedural complications) | 0 | 1
Burn (Injury, poisoning and procedural complications) | 1 | 1
Bruising (Injury, poisoning and procedural complications) | 6 | 8
Ankle Fracture (Injury, poisoning and procedural complications) | 2 | 0
Investigations - Other (Investigations) | 2 | 4
Weight Loss (Investigations) | 19 | 25
Weight Gain (Investigations) | 5 | 4
Platelet Count Decreased (Investigations) | 30 | 18
Lymphocyte Count Decreased (Investigations) | 10 | 15
Inr Increased (Investigations) | 5 | 3
Hemoglobin Increased (Investigations) | 1 | 0
Ggt Increased (Investigations) | 2 | 2
Electrocardiogram Qt Corrected Interval Prolonged (Investigations) | 1 | 0
Ejection Fraction Decreased (Investigations) | 1 | 3
Creatinine Increased (Investigations) | 9 | 11
Cholesterol High (Investigations) | 1 | 1
Neutrophil Count Decreased (Investigations) | 60 | 54
Urine Output Decreased (Investigations) | 1 | 0
Cd4 Lymphocytes Decreased (Investigations) | 1 | 2
Blood Bilirubin Increased (Investigations) | 1 | 0
White Blood Cell Decreased (Investigations) | 83 | 74
Aspartate Aminotransferase Increased (Investigations) | 14 | 17
Alkaline Phosphatase Increased (Investigations) | 18 | 18
Alanine Aminotransferase Increased (Investigations) | 12 | 9
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1 | 1
Metabolism And Nutrition Disorders - Other (Metabolism and nutrition disorders) | 3 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 10 | 6
Hyponatremia (Metabolism and nutrition disorders) | 18 | 21
Hypomagnesemia (Metabolism and nutrition disorders) | 28 | 24
Hypokalemia (Metabolism and nutrition disorders) | 28 | 12
Hypoglycemia (Metabolism and nutrition disorders) | 7 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 14 | 15
Hypoalbuminemia (Metabolism and nutrition disorders) | 27 | 23
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 2
Hypernatremia (Metabolism and nutrition disorders) | 5 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 8 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 28 | 19
Hypercalcemia (Metabolism and nutrition disorders) | 3 | 3
Glucose Intolerance (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 9 | 11
Anorexia (Metabolism and nutrition disorders) | 46 | 48
Alkalosis (Metabolism and nutrition disorders) | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 15 | 23
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 24 | 20
Muscle Weakness Upper Limb (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscle Weakness Left-Sided (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 12 | 16
Flank Pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Buttock Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 8 | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 26 | 30
Avascular Necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 17
Abdominal Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal And Connective Tissue Disorder - (Musculoskeletal and connective tissue disorders) | 4 | 2
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nervous System Disorders - Other (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 3 | 3
Transient Ischemic Attacks (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 47 | 45
Peripheral Motor Neuropathy (Nervous system disorders) | 6 | 5
Paresthesia (Nervous system disorders) | 5 | 7
Neuralgia (Nervous system disorders) | 2 | 0
Memory Impairment (Nervous system disorders) | 3 | 2
Lethargy (Nervous system disorders) | 0 | 1
Hypersomnia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 34 | 27
Facial Nerve Disorder (Nervous system disorders) | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 13 | 7
Dysarthria (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 14 | 24
Depressed Level Of Consciousness (Nervous system disorders) | 0 | 1
Concentration Impairment (Nervous system disorders) | 0 | 1
Cognitive Disturbance (Nervous system disorders) | 1 | 3
Ataxia (Nervous system disorders) | 1 | 1
Akathisia (Nervous system disorders) | 0 | 1
Psychiatric Disorders - Other (Psychiatric disorders) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 0 | 2
Psychosis (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 16 | 27
Hallucinations (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 24 | 24
Confusion (Psychiatric disorders) | 4 | 6
Anxiety (Psychiatric disorders) | 24 | 32
Agitation (Psychiatric disorders) | 1 | 6
Renal And Urinary Disorders - Other (Renal and urinary disorders) | 2 | 6
Urine Discoloration (Renal and urinary disorders) | 1 | 0
Urinary Urgency (Renal and urinary disorders) | 2 | 5
Urinary Tract Obstruction (Renal and urinary disorders) | 5 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 5 | 11
Urinary Tract Pain (Renal and urinary disorders) | 4 | 1
Urinary Frequency (Renal and urinary disorders) | 7 | 13
Proteinuria (Renal and urinary disorders) | 3 | 1
Hemoglobinuria (Renal and urinary disorders) | 2 | 0
Hematuria (Renal and urinary disorders) | 5 | 1
Chronic Kidney Disease (Renal and urinary disorders) | 3 | 3
Acute Kidney Injury (Renal and urinary disorders) | 1 | 2
Reproductive System And Breast Disorders - Other (Reproductive system and breast disorders) | 0 | 1
Vaginal Pain (Reproductive system and breast disorders) | 1 | 0
Vaginal Hemorrhage (Reproductive system and breast disorders) | 6 | 5
Vaginal Dryness (Reproductive system and breast disorders) | 3 | 1
Pelvic Pain (Reproductive system and breast disorders) | 4 | 5
Vaginal Discharge (Reproductive system and breast disorders) | 8 | 5
Vaginal Inflammation (Reproductive system and breast disorders) | 1 | 1
Breast Pain (Reproductive system and breast disorders) | 1 | 0
Respiratory, Thoracic And Mediastinal Disorders - (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal Mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 40 | 39
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 36
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 8 | 15
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 3
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Ulceration (Skin and subcutaneous tissue disorders) | 4 | 5
Skin Induration (Skin and subcutaneous tissue disorders) | 1 | 7
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 20 | 21
Scalp Pain (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 7 | 9
Purpura (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 24 | 20
Photosensitivity (Skin and subcutaneous tissue disorders) | 2 | 1
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 55 | 54
Pain Of Skin (Skin and subcutaneous tissue disorders) | 6 | 4
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 58 | 53
Nail Ridging (Skin and subcutaneous tissue disorders) | 1 | 2
Nail Loss (Skin and subcutaneous tissue disorders) | 2 | 2
Nail Discoloration (Skin and subcutaneous tissue disorders) | 8 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 3
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 5 | 8
Dry Skin (Skin and subcutaneous tissue disorders) | 21 | 24
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 6 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 14 | 20
Surgical And Medical Procedures - Other (Surgical and medical procedures) | 1 | 3
Vascular Disorders - Other (Vascular disorders) | 1 | 0
Thromboembolic Event (Vascular disorders) | 7 | 5
Superficial Thrombophlebitis (Vascular disorders) | 1 | 0
Lymphedema (Vascular disorders) | 5 | 4
Hypotension (Vascular disorders) | 6 | 11
Hypertension (Vascular disorders) | 13 | 18
Hot Flashes (Vascular disorders) | 13 | 7
Hematoma (Vascular disorders) | 3 | 4
Flushing (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No